CLINICAL TRIAL: NCT00968890
Title: Immunogenicity, Safety and Reactogenicity of GSK Biologicals' Influenza GSK2340272A and Fluarix™ 2009-2010 Vaccines When Co-administered in Elderly Subjects Aged 61 Years and Older
Brief Title: Immunogenicity and Safety of Vaccine GSK2340272A (H1N1) and GSK Biologicals Fluarix™ Vaccine When Co-administered in Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113525
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Results first posted 2011-03-16 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340272A; Influenza infection
MeSH Terms: conditions — Influenza, Human | interventions — pandemrix; fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Pandemrix+Fluarix and Pandemrix+Placebo (Experimental): Subjects received two doses of Pandemrix (GSK2340272A) intramuscularly in the deltoid region of the non-dominant arm co-administered with Fluarix™ on Day 0 and with a placebo on Day 21 intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: Pandemrix (Influenza vaccine GSK2340272A); Biological: Fluarix™; Biological: Placebo
- Pandemrix+Placebo and Pandemrix+Fluarix (Experimental): Subjects received two doses of Pandemrix (GSK2340272A) intramuscularly in the deltoid region of the non-dominant arm co-administered with a placebo on Day 0 and with Fluarix™ on Day 21 intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: Pandemrix (Influenza vaccine GSK2340272A); Biological: Fluarix™; Biological: Placebo

INTERVENTIONS:
Biological: Pandemrix (Influenza vaccine GSK2340272A) — Intramuscular injection, 2 doses
Biological: Fluarix™ — Intramuscular injection, 1 dose
  Other Names: 2009-2010 Northern Hemisphere trivalent seasonal influenza vaccine
Biological: Placebo — Intramuscular injection, 1 dose

SUMMARY:
The purpose of the present study is to assess the immunogenicity, safety and reactogenicity of a two-dose schedule with vaccine GSK2340272A when co-administered with GSK Biologicals' Fluarix™ vaccine either at the time of first or second vaccination in elderly subjects aged 61 years and older.

DETAILED DESCRIPTION:
The study will be conducted in an open manner regarding the administration of vaccine GSK2340272A.

The study will be observer-blind regarding the administration of Fluarix™ and placebo vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 61 years of age or older at the time of the first vaccination
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination.
* Access to a consistent means of telephone contact.

Exclusion Criteria:

* Previous administration of the 2009 Southern Hemisphere or 2009-2010 Northern Hemisphere seasonal influenza vaccine.
* Previous administration of a pandemic influenza vaccine.
* Administration of any vaccine within 30 days before first vaccination.
* Planned administration of a vaccine not foreseen by the study protocol one month (minimum 30 days) after the second vaccination with vaccine GSK2340272A.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of the study vaccines or planned use during the study period. Potential subjects in the follow-up (i.e., no treatment) phase of a prior investigational study may be enrolled if the investigator's judgment is that it will have no effect on safety, reactogenicity, or immunogenicity endpoints in this study, and that it does not violate the protocol requirements of the prior trial.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an oral temperature >= 37.5°C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Chronic administration of immunosuppressants or other immune modifying drugs within six months prior to the first vaccination.
* Receipt of any immunoglobulins and/or any blood products within 3 months preceding the first vaccination or planned administration of any of these products during the entire study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic anti-platelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Serious chronic disease as determined by medical history and physical examination.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormalities, as determined by physical examination or laboratory screening tests.
* Any known or suspected allergy to any constituent of influenza vaccines.
* History of chronic alcohol consumption and/or drug abuse.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Min Age: 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-09-12; Primary Completion 2010-09-23 (Actual); Study Completion 2010-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Sweden (2):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Örebro

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Peeters M, Regner S, Vaman T, Devaster JM, Rombo L. Safety and immunogenicity of an AS03-adjuvanted A(H1N1)pmd09 vaccine administered simultaneously or sequentially with a seasonal trivalent vaccine in adults 61 years or older: data from two multicentre randomised trials. Vaccine. 2012 Oct 5;30(45):6483-91. doi: 10.1016/j.vaccine.2012.07.081. Epub 2012 Aug 9. PMID 22885014
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 113525 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113525 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113525 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113525 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113525 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113525 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113525 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Started | 84 | 84
Completed | 84 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.9 (4.63) | 69.1 (4.70) | 69.0 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 89
  Male | 42 | 37 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects After the Second Dose of Pandemrix and After Vaccination With Fluarix
Description: A seroconverted subject is a subject who had either a pre-vaccination reciprocal hemagglutination inhibition (HI) titer < 10 and a postvaccination reciprocal titer >= 40, or a pre-vaccination reciprocal HI titer >= 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus.
  The Pandemrix vaccine strain was A/Cal/09. The Fluarix vaccine strains were A/Bri/07, A/Uru/07 and B/Bri/08.
Time Frame: 21 days after the second dose of Pandemrix (=Day 42) and after vaccination with Fluarix (=Day 21 for Pandemrix+Fluarix and Pandemrix+Placebo Group or Day 42 for Pandemrix+ Placebo and Pandemrix+Fluarix Group)
Population: The analysis was performed on the according-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom blood samples were taken and immunogenicity data were available.
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 83 | 84
subjects
  A/Cal/09 | 79 | 82
  B/Bri/08 | 40 | 22
  A/Uru/07 | 36 | 23
  A/Bri/07 | 31 | 23

2. Primary Outcome: Number of Seroprotected Subjects After the Second Dose of Pandemrix and After Vaccination With Fluarix
Description: A seroprotected subject was a subject with reciprocal HI titers >= 40 against the vaccine homologous virus.
  The Pandemrix vaccine strain was A/Cal/09. The Fluarix vaccine strains were A/Bri/07, A/Uru/07 and B/Bri/08.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 83 | 84
subjects
  A/Cal/09 | 82 | 84
  A/Bri/07 | 57 | 52
  A/Uru/07 | 65 | 54
  B/Bri/08 | 83 | 84

3. Primary Outcome: Geometric Mean Fold Rise (GMFR) After the Second Dose of Pandemrix and After Vaccination With Fluarix
Description: The GMFR is defined as the Geometric Mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus.
  The Pandemrix vaccine strain was A/Cal/09. The Fluarix vaccine strains were A/Bri/07, A/Uru/07 and B/Bri/08.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 83 | 84
ratio
  A/Cal/09 | 33.1 [26.0 to 42.1] | 32.2 [25.6 to 40.4]
  B/Bri/08 | 4.7 [3.6 to 6.1] | 2.1 [1.8 to 2.5]
  A/Uru/07 | 4.2 [3.3 to 5.4] | 3.0 [2.4 to 3.9]
  A/Bri/07 | 3.5 [2.9 to 4.3] | 2.7 [2.2 to 3.3]

4. Secondary Outcome: Geometric Mean Titers for Antibodies Against Pandemrix and Fluarix Vaccine Strains
Description: Titers are expressed as GMTs.
  The Pandemrix vaccine strain was A/Cal/09. The Fluarix vaccine strains were A/Bri/07, A/Uru/07 and B/Bri/08.
Time Frame: Days 0, 21, 42, 182, 364
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
titer
  A/Cal/09 Day 0 (N=83;84) | 7.4 [6.1 to 9.0] | 8.5 [7.1 to 10.2]
  A/Cal/09 Day 21 (N=83;84) | 138.8 [107.7 to 178.9] | 168.2 [137.5 to 205.7]
  A/Cal/09 Day 42 (N=83;84) | 246.1 [201.3 to 300.8] | 273.6 [231.4 to 323.4]
  A/Cal/09 Day 182 (N=84;84) | 71.2 [57.4 to 88.4] | 84.0 [69.8 to 101.2]
  A/Cal/09 Day 364 (N=84;84) | 29.1 [22.8 to 37.0] | 34.4 [28.0 to 42.4]
  A/Bri/07 Day 0 (N=83;84) | 15.2 [12.4 to 18.7] | 16.0 [13.3 to 19.2]
  A/Bri/07 Day 21/Day 42 (N=83;84) | 53.6 [43.1 to 66.5] | 42.5 [34.5 to 52.4]
  A/Bri/07 Day 182 (N=84;84) | 37.9 [31.6 to 45.4] | 36.8 [30.5 to 44.4]
  A/Bri/07 Day 364 (N=84;84) | 29.4 [24.9 to 34.7] | 28.8 [24.4 to 34.0]
  A/Uru/07 Day 0 (N=83;84) | 17.9 [14.0 to 22.8] | 19.7 [15.0 to 25.8]
  A/Uru/07 Day 21/Day 42 (N=83;84) | 74.8 [57.6 to 97.1] | 59.7 [44.5 to 80.0]
  A/Uru/07 Day 182 (N=84;84) | 35.9 [28.0 to 46.0] | 35.0 [26.2 to 46.9]
  A/Uru/07 Day 364 (N=84;84) | 28.7 [22.8 to 36.3] | 27.7 [20.6 to 37.2]
  B/Bri/08 Day 0 (N=83;84) | 49.9 [38.8 to 64.1] | 115.5 [96.3 to 138.5]
  B/Bri/08 Day 21/Day 42 (N=83;84) | 235.0 [199.5 to 276.8] | 246.7 [208.5 to 292.0]
  B/Bri/08 Day 182 (N=84;84) | 220.7 [187.9 to 259.3] | 222.5 [188.6 to 262.6]
  B/Bri/08 Day 364 (N=84;84) | 104.6 [88.5 to 123.7] | 112.7 [92.4 to 137.4]

5. Secondary Outcome: Number of Seroconverted Subjects
Description: as for outcome 1
Time Frame: at Day 21 (for Pandemrix vaccine strain only), Day 182 and Day 364
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
subjects
  A/Cal/09 Day 21 (N=83;84) | 73 | 78
  A/Cal/09 Day 182 (N=84;84) | 64 | 69
  A/Cal/09 Day 364 (N=84;84) | 25 | 30
  A/Bri/07 Day 182 (N=84;84) | 18 | 13
  A/Bri/07 Day 364 (N=84;84) | 5 | 8
  A/Uru/07 Day 182 (N=84;84) | 13 | 9
  A/Uru/07 Day 364 (N=84;84) | 7 | 6
  B/Bri/08 Day 182 (N=84;84) | 40 | 13
  B/Bri/08 Day 364 (N=84;84) | 19 | 3

6. Secondary Outcome: Number of Seroprotected Subjects
Description: A seroprotected subject is a subject with reciprocal HI titers >= 40 against the vaccine homologous virus. The Pandemrix vaccine strain was A/Cal/09. The Fluarix vaccine strains were A/Bri/07, A/Uru/07 and B/Bri/08.
Time Frame: at Day 21 (for Pandemrix vaccine strain only), Day 182 and Day 364
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
subjects
  A/Cal/09 Day 0 (N=83;84) | 6 | 7
  A/Cal/09 Day 21 (N=83;84) | 74 | 81
  A/Cal/09 Day 182 (N=84;84) | 67 | 75
  A/Cal/09 Day 364 (N=84;84) | 32 | 40
  A/Bri/07 Day 0 (N=83;84) | 22 | 17
  A/Bri/07 Day 182 (N=84;84) | 48 | 44
  A/Bri/07 Day 364 (N=84;84) | 36 | 34
  A/Uru/07 Day 0 (N=83;84) | 29 | 31
  A/Uru/07 Day 182 (N=84;84) | 44 | 43
  A/Uru/07 Day 364 (N=84;84) | 36 | 40
  B/Bri/08 Day 0 (N=83;84) | 56 | 78
  B/Bri/08 Day 182 (N=84;84) | 84 | 84
  B/Bri/08 Day 364 (N=84;84) | 78 | 77

7. Secondary Outcome: Geometric Mean Fold Rise (GMFR)
Description: as for outcome 3
Time Frame: at Day 21 (for Pandemrix vaccine strain only), Day 182 and Day 364
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
ratio
  A/Cal/09 Day 21 (N=83;84) | 18.7 [14.6 to 23.8] | 19.8 [15.7 to 25.0]
  A/Cal/09 Day 182 (N=84;84) | 9.6 [7.8 to 11.9] | 9.9 [8.1 to 12.0]
  A/Cal/09 Day 364 (N=84;84) | 3.9 [3.2 to 4.8] | 4.0 [3.3 to 4.9]
  A/Bri/07 Day 182 (N=84;84) | 2.5 [2.1 to 2.9] | 2.3 [2.0 to 2.7]
  A/Bri/07 Day 364 (N=84;84) | 1.9 [1.7 to 2.2] | 1.8 [1.6 to 2.1]
  A/Uru/07 Day 182 (N=84;84) | 2.0 [1.6 to 2.4] | 1.8 [1.5 to 2.1]
  A/Uru/07 Day 364 (N=84;84) | 1.6 [1.4 to 1.9] | 1.4 [1.2 to 1.7]
  B/Bri/08 Day 182 (N=84;84) | 4.4 [3.6 to 5.5] | 1.9 [1.7 to 2.2]
  B/Bri/08 Day 364 (N=84;84) | 2.1 [1.7 to 2.6] | 1.0 [0.9 to 1.0]

8. Secondary Outcome: Number of Subjects With Titers Equal to or Above Titer 1:10
Description: The cut-off 1:10 was considered as seropositivity.
  The Pandemrix vaccine strain was A/Cal/09. The Fluarix vaccine strains were A/Bri/07, A/Uru/07 and B/Bri/08.
Time Frame: Days 0, 21, 42, 182, 364
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
subjects
  A/Cal/09 Day 0 (N=83;84) | 20 | 32
  A/Cal/09 Day 21 (N=83;84) | 82 | 84
  A/Cal/09 Day 42 (N=83;84) | 83 | 84
  A/Cal/09 Day 182 (N=84;84) | 84 | 84
  A/Cal/09 Day 364 (N=84;84) | 78 | 81
  A/Bri/07 Day 0 (N=83;84) | 59 | 68
  A/Bri/07 Day 21/Day 42 (N=83;84) | 82 | 82
  A/Bri/07 Day 182 (N=84;84) | 83 | 83
  A/Bri/07 Day 364 (N=84;84) | 82 | 83
  A/Uru/07 Day 0 (N=83;84) | 58 | 57
  A/Uru/07 Day 21/Day 42 (N=83;84) | 79 | 80
  A/Uru/07 Day 182 (N=84;84) | 77 | 73
  A/Uru/07 Day 364 (N=84;84) | 76 | 65
  B/Bri/08 Day 0 (N=83;84) | 76 | 84
  B/Bri/08 Day 21/Day 42 (N=83;84) | 83 | 84
  B/Bri/08 Day 182 (N=84;84) | 84 | 84
  B/Bri/08 Day 364 (N=84;84) | 84 | 84

9. Secondary Outcome: Number of Subjects With Solicited Local and General Symptoms
Description: Solicited local symptoms are pain, redness and swelling at the injection site. They are divided between solicited local symptoms occurring after administration of Pandemrix, Fluarix or Placebo. Solicited general symptoms are fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and temperature (defined as axillary temperature >= 38.0 degrees Celsius).
Time Frame: Within 7 days (Day 0-Day 6) after each vaccination
Population: Analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
subjects
  Pain after Pandemrix | 64 | 74
  Pain after Fluarix | 18 | 26
  Pain after Placebo | 0 | 8
  Redness after Pandemrix | 15 | 19
  Redness after Fluarix | 0 | 1
  Redness after Placebo | 0 | 0
  Swelling after Pandemrix | 22 | 27
  Swelling after Fluarix | 3 | 4
  Swelling after Placebo | 0 | 2
  Fatigue | 25 | 27
  Headache | 23 | 23
  Joint pain at other location | 13 | 17
  Muscle aches | 18 | 26
  Shivering | 12 | 16
  Sweating | 2 | 8
  Temperature | 3 | 0

10. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms
Time Frame: From Day 0 to Day 83
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
subjects | 41 | 41

11. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest
Description: Adverse events of specific interest include autoimmune diseases and other immune mediated inflammatory disorders.
Time Frame: From Day 0 to Day 364
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
subjects | 0 | 0

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to Day 364
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Number analyzed (Participants) | 84 | 84
subjects | 2 | 3

ADVERSE EVENTS:
Arm/Group | Pandemrix+Fluarix and Pandemrix+Placebo | Pandemrix+Placebo and Pandemrix+Fluarix
Serious Adverse Events (participants affected / at risk) | 2/84 | 3/84
Other Adverse Events (participants affected / at risk) | 71/84 | 78/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pandemrix+Fluarix and Pandemrix+Placebo (N=84) | Pandemrix+Placebo and Pandemrix+Fluarix (N=84)
Cardiac failure (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pandemrix+Fluarix and Pandemrix+Placebo (N=84) | Pandemrix+Placebo and Pandemrix+Fluarix (N=84)
Pain after Pandemrix (General disorders) | 64 | 74
Pain after Fluarix (General disorders) | 18 | 26
Pain after Placebo (General disorders) | 0 | 8
Redness after Pandemrix (General disorders) | 15 | 19
Swelling after Pandemrix (General disorders) | 22 | 27
Fatigue (General disorders) | 25 | 27
Headache (General disorders) | 23 | 23
Joint pain at other location (General disorders) | 13 | 17
Muscle aches (General disorders) | 18 | 26
Shivering (General disorders) | 12 | 16
Sweating (General disorders) | 2 | 8
Nasopharyngitis (Infections and infestations) | 15 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 2 | 5
Dizziness (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.